CLINICAL TRIAL: NCT05777343
Title: Pain Neuroscience Education, Exercise, and Cognitive Training in Individuals With Idiopathic Chronic Low Back Pain: a Three-arm Randomized Trial
Brief Title: Exercise, PNE and Cognitive Training in Individuals With Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aveiro University (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other); RISE Study Group (Network)
Responsible Party: Principal Investigator, Ellen Hirose Pereira Nery, Principal Investigator, Aveiro University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCTCognitiveTraining
Record Dates: First submitted 2023-02-23; First posted 2023-03-21 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Chronic Low-back Pain
Keywords: cognitive training; exercise; chronic low back pain; pain neuroscience education
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention 1 (Experimental): Participants will receive exercise, PNE and online cognitive training sessions.
  Interventions: Other: Experimental
- Intervention 2 (Active Comparator): Participants will receive exercise and pain neuroscience education (PNE).
  Interventions: Other: Exercise and PNE
- Intervention 3 (Active Comparator): Participants will receive online cognitive training sessions.
  Interventions: Other: Cognitive training

INTERVENTIONS:
Other: Experimental — Cognitive training combined with the recommended non-pharmacological intervention (Exercise and Pain Neuroscience Education).
  Arms: Intervention 1
Other: Exercise and PNE — Recommended non-pharmacological intervention (Exercise and Pain Neuroscience Education).
  Arms: Intervention 2
Other: Cognitive training — Online sessions of cognitive training.
  Arms: Intervention 3

SUMMARY:
This study aims of to investigate whether combining cognitive training to exercise and Pain Neuroscience Education will contribute to reduction of pain and associated symptoms (i.e., catastrophizing, fear of movement, disability) in individuals with low back pain (LBP).

DETAILED DESCRIPTION:
This study aims of to investigate whether combining cognitive training to exercise and Pain Neuroscience Education (PNE) will contribute to reduction of pain and associated symptoms (i.e., catastrophizing, fear of movement, disability) in individuals with low back pain (LBP).

It will have three arms of which will receive exercise, PNE and/or cognitive training for 8 weeks (Group I - exercise and PNE; Group II - exercise, PNE and cognitive training; Group III - cognitive training).

Participants will be assessed for pain characteristics, psychological, and cognitive aspects at baseline, post-intervention and at 3 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* have chronic idiopathic LBP
* report pain intensity of at least 2 out of 10 on the Numeric Pain Rating Scale
* 18 to 64 years old
* Be able to read, write and speak Portuguese
* Asses to personal computer and internet for those receiving cognitive training

Exclusion Criteria:

* individuals receiving any chronic treatment for their pain
* symptoms of peripheral nervous system pathology (e.g., motor weakness and sensory disturbance);
* a diagnosis of an ongoing neurological disease with peripheral or central nervous system involvement or relevant sequela;
* having a diagnosis of ongoing psychiatric disease
* having relevant cognitive impairment as assessed by Montreal Cognitive Assessment (MoCA).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-02-10 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale Numeric Pain Rating Scale | baseline
  Measured with a 11-point scale ranging from 0 meaning "no pain" to 10 meaning "the worst pain imaginable".
Numeric Pain Rating Scale Numeric Pain Rating Scale | post-intervention - 8 weeks
  Measured with a 11-point scale ranging from 0 meaning "no pain" to 10 meaning "the worst pain imaginable".
Numeric Pain Rating Scale Numeric Pain Rating Scale | 3 months follow-up
  Measured with a 11-point scale ranging from 0 meaning "no pain" to 10 meaning "the worst pain imaginable".

SECONDARY OUTCOMES:
Cognitive Function | baseline
  Cognitive function will be assessed using the Brain on Track® (BoT), a self-administered computerized test that evaluates different cognitive domains. Each test has a virtually unlimited range score and considers the maximum number of correct answers that a person gives in a fixed period of time and higher scores represent higher cognitive performance.
Cognitive Function | post-intervention - 8 weeks
  Cognitive function will be assessed using the Brain on Track® (BoT), a self-administered computerized test that evaluates different cognitive domains. Each test has a virtually unlimited range score and considers the maximum number of correct answers that a person gives in a fixed period of time and higher scores represent higher cognitive performance.
Cognitive Function | 3 months follow-up.
  Cognitive function will be assessed using the Brain on Track® (BoT), a self-administered computerized test that evaluates different cognitive domains. Each test has a virtually unlimited range score and considers the maximum number of correct answers that a person gives in a fixed period of time and higher scores represent higher cognitive performance.
Roland Morris disability questionnaire | baseline
  The Roland Morris assesses disability caused by LBP. It has 24 statements, and the individual must tick those that relate to him that day. The total score ranges from "0" meaning no disability to "24" meaning maximum disability.
Roland Morris disability questionnaire | post-intervention - 8 weeks
  The Roland Morris assesses disability caused by LBP. It has 24 statements, and the individual must tick those that relate to him that day. The total score ranges from "0" meaning no disability to "24" meaning maximum disability.
Roland Morris disability questionnaire | 3 months follow-up
  The Roland Morris assesses disability caused by LBP. It has 24 statements, and the individual must tick those that relate to him that day. The total score ranges from "0" meaning no disability to "24" meaning maximum disability.
Central sensitization Inventory | baseline
  The central sensitization inventory (CSI) assesses symptoms of central sensitization. The total score ranges from 0 to 100 points and to identify central sensitization in individuals, the recommended cut-off score is 40 points.
Central sensitization Inventory | post-intervention - 8 weeks
  The central sensitization inventory (CSI) assesses symptoms of central sensitization. The total score ranges from 0 to 100 points and to identify central sensitization in individuals, the recommended cut-off score is 40 points.
Central sensitization Inventory | 3 months follow-up
  The central sensitization inventory (CSI)assesses symptoms of central sensitization. The total score ranges from 0 to 100 points and to identify central sensitization in individuals, the recommended cut-off score is 40 points.
Hospital Anxiety and Depression Scale (HADS) | baseline
  HADS evaluates symptoms of anxiety and depression. The total scores range from 0 to 21 points with a 4-point Likert scale rating between "most of the times" and "not at all" with higher scores indicating higher levels of anxiety and depression.
Hospital Anxiety and Depression Scale (HADS) | post-intervention - 8 weeks
  HADS evaluates symptoms of anxiety and depression. The total scores range from 0 to 21 points with a 4-point Likert scale rating between "most of the times" and "not at all" with higher scores indicating higher levels of anxiety and depression.
Hospital Anxiety and Depression Scale (HADS) | 3 months follow-up.
  HADS evaluates symptoms of anxiety and depression. The total scores range from 0 to 21 points with a 4-point Likert scale rating between "most of the times" and "not at all" with higher scores indicating higher levels of anxiety and depression.
TAMPA Scale of Kinesiophobia | baseline
  The Tampa scale measures the fear of movement related to chronic LBP. The short version has 13 items in a 4-point Likert scale rating between "strongly disagree" and "strongly agree". The total scores range from 0 to 52 points with higher levels indicating higher fear of movement.
TAMPA Scale of Kinesiophobia | post-intervention - 8 weeks
  The Tampa scale measures the fear of movement related to chronic LBP. The short version has 13 items in a 4-point Likert scale rating between "strongly disagree" and "strongly agree". The total scores range from 0 to 52 points with higher levels indicating higher fear of movement.
TAMPA Scale of Kinesiophobia | 3 months follow-up.
  The Tampa scale measures the fear of movement related to chronic LBP. The short version has 13 items in a 4-point Likert scale rating between "strongly disagree" and "strongly agree". The total scores range from 0 to 52 points with higher levels indicating higher fear of movement.
Pain Catastrophizing Scale | Baseline
  The Pain Catastrophizing Scale (PCS) assess catastrophic thinking related to pain. It has 13 statements on a 5-point scale ranging from 0 meaning "not at all" and 4 meaning "all the time". The total score ranges from 0 to 52 with higher scores indicating higher levels of catastrophizing.
Pain Catastrophizing Scale | post-intervention - 8 weeks
  The Pain Catastrophizing Scale (PCS) assess catastrophic thinking related to pain. It has 13 statements on a 5-point scale ranging from 0 meaning "not at all" and 4 meaning "all the time". The total score ranges from 0 to 52 with higher scores indicating higher levels of catastrophizing.
Pain Catastrophizing Scale | 3 months follow-up.
  The Pain Catastrophizing Scale (PCS) assess catastrophic thinking related to pain. It has 13 statements on a 5-point scale ranging from 0 meaning "not at all" and 4 meaning "all the time". The total score ranges from 0 to 52 with higher scores indicating higher levels of catastrophizing.
Basic Scale on Insomnia Complaints and Quality of Sleep (BaSIQs) | baseline
  The scale assess the difficulties with sleep onset and maintenance and the quality and depth of sleep during the last month and considering a normal week. Total score ranges from 0 to 28 points and higher scores are associated with poor quality of sleep.
Basic Scale on Insomnia Complaints and Quality of Sleep (BaSIQs) | post-intervention - 8 weeks
  The scale assess the difficulties with sleep onset and maintenance and the quality and depth of sleep during the last month and considering a normal week. Total score ranges from 0 to 28 points and higher scores are associated with poor quality of sleep.
Basic Scale on Insomnia Complaints and Quality of Sleep (BaSIQs) | 3 months follow-up.
  The scale assess the difficulties with sleep onset and maintenance and the quality and depth of sleep during the last month and considering a normal week. Total score ranges from 0 to 28 points and higher scores are associated with poor quality of sleep.
Two-point discrimination | baseline
  Two-point discrimination is used to assess cortical reorganization.
Two-point discrimination | post-intervention - 8 weeks
  Two-point discrimination is used to assess cortical reorganization.
Two-point discrimination | 3 months follow-up
  Two-point discrimination is used to assess cortical reorganization.
Patient's Global Impression of Change (PGIC) | post-intervention - 8 weeks
  PGIC evaluates the perception of improvement associated with the intervention. Participants are instructed to select on a scale from 1 ("No change or condition worsened") to 7 ("Much better, and with a considerable improvement that made all the difference") the statement that best reflected the impact of the intervention on their condition.
Patient's Global Impression of Change (PGIC) | 3 months follow-up.
  PGIC evaluates the perception of improvement associated with the intervention. Participants are instructed to select on a scale from 1 ("No change or condition worsened") to 7 ("Much better, and with a considerable improvement that made all the difference") the statement that best reflected the impact of the intervention on their condition.

CONTACTS AND LOCATIONS:
Overall Officials: Anabela Silva, PhD, Study Director — School of Health Sciences, University of Aveiro
Locations (1):
- University of Aveiro, Aveiro, Portugal